CLINICAL TRIAL: NCT06392516
Title: Effect of Intradialytic Administration of Ketoacid Analogues on Inflammatory Parameters in Patients Undergoing Chronic Hemodialysis Twice a Week
Brief Title: Ketoacid Analogues Intradialytic Effect on Inflammation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RSUP Fatmawati (Other)
Responsible Party: Principal Investigator, Anggraini Permata Sari, Internal Medicine Staff, Fellow of Nephrology Division, RSUP Fatmawati
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RSF_IPDGH_01
Record Dates: First submitted 2024-04-23; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Hemodialysis Complication
Keywords: ketoacid analogues; inflammation; hemodialysis
MeSH Terms: conditions — Inflammation | interventions — Keto Acids

STUDY DESIGN:
Intervention Model Description: intervention and control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (No Intervention): patient who undergo hemodialysis two times a week
- intervention (Experimental): will be given parenteral ketoacid analogues intradialytics two times a week
  Interventions: Drug: Ketoacid

INTERVENTIONS:
Drug: Ketoacid — 250 ml ketoacid two hours before the hemodialysis session ended
  Arms: intervention

SUMMARY:
this study tries to measure the effect of intradialytic ketoacid analogues on inflammatory parameters

DETAILED DESCRIPTION:
this study will measure inflammation parameters:

* interleukin 6
* malnutrition inflammation score
* neutrophil lymphocyte ratio
* monocyte lymphocyte ratio
* thrombocyte lymphocyte ratio

the duration of intervention is 12 weeks

ELIGIBILITY:
Inclusion Criteria:

* patient who undergo hemodialysis two times a week

Exclusion Criteria:

* travelling hemodialysis
* acute conditions
* HIV patient
* acute infection
* stroke and immobilized patient

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2024-04-29 (Estimated); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
interleukin-6 | 12 weeks
  in pg/mL, no limit values
malnutrition inflammation score | 12 weeks
  consists of ten components, based on subjective complaints combined with albumin serum (in g/dL), serum iron (in micromol/L, and total iron binding capacity (in micromol/L). the sum of all components >5 means have high inflammation status
neutrophil lymphocyte ratio | 12 weeks
  the percentage ratio of neutrophil count and lymphocyte count will be combined to neutrophil lymphocyte ratio
monocyte lymphocyte ratio | 12 weeks
  the percentage ratio of monocyte count and lymphocyte count will be combined to monocyte lymphocyte ratio
thrombocyte lymphocyte ratio | 12 weeks
  the percentage ratio of thrombocyte (in per microliter of blood) and lymphocyte count will be combined to thrombocyte lymphocyte ratio

CONTACTS AND LOCATIONS:
Locations (1):
- RSUP Fatmawati, Jakarta, Jakarta Selatan, Indonesia

IPD SHARING:
Plan to Share IPD: No
the data is restricted only for investigators